CLINICAL TRIAL: NCT05731596
Title: Comparative Clinical Study to Evaluate the Possible Efficacy and Safety of Rosuvastatin Versus Coenzyme Q10 on Nonalcoholic Steatohepatitis
Brief Title: Comparative Clinical Study to Evaluate the Efficacy and Safety of Rosuvastatin Vs CoQ10 on Nonalcoholic Steatohepatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hadeer Ahmed Alsayed, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rosuvastatin vs Co Q10 on NASH
Record Dates: First submitted 2023-01-16; First posted 2023-02-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: nonalcoholic steatohepatitis; NASH; NAFLD; Non-Alcoholic Fatty Liver Disease; Rosuvastatin; Coenzyme Q10; Fatty Liver; statin; Liver Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases | interventions — Rosuvastatin Calcium; Tablets; coenzyme Q10

STUDY DESIGN:
Intervention Model Description: * This study will be a randomized, controlled, parallel study.
  * It will be conducted on 46 patients diagnosed with NASH
  * The patients will be randomized into two groups:
    1. Group 1(n=23): patients will receive Rosuvastatin 20mg/day orally
    2. Group 2(n=23): patients will receive Coenzyme Q10 100 mg/day orally
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Rosuvastatin group) (Active Comparator): Patients will receive Rosuvastatin 20mg/day orally for 3 months
  Interventions: Drug: Rosuvastatin 20 Mg Oral Tablet
- Group 2 (CoQ10 group) (Experimental): Patients will receive Coenzyme Q10 100 mg/day orally for 3 months
  Interventions: Drug: Coenzyme Q10 100 MG Oral Capsule

INTERVENTIONS:
Drug: Rosuvastatin 20 Mg Oral Tablet — Rosuvastatin 20 mg will be administered orally once daily for 3 Months
  Arms: Group 1 (Rosuvastatin group)
Drug: Coenzyme Q10 100 MG Oral Capsule — Coenzyme Q10 100 mg will be administered orally once daily for 3 Months
  Arms: Group 2 (CoQ10 group)

SUMMARY:
This study will be a randomized, controlled, parallel study that aims to evaluate the efficacy and safety of Rosuvastatin versus Coenzyme Q10 on nonalcoholic steatohepatitis patients.

DETAILED DESCRIPTION:
* This study will be a randomized, controlled, parallel study.
* It will be conducted on 46 patients diagnosed with NASH
* The patients will be randomized into two groups:

Group 1(n=23): patients will receive Rosuvastatin 20mg/day orally

Group 2(n=23): patients will receive Coenzyme Q10 100 mg/day orally

The patients will be selected from community awareness campaigns about NASH in Alexandria , Egypt . Written informed consent will be obtained from all patients. This study will be approved by the Research Ethics Committee of Tanta University and Alexandria university.

The study duration will be 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years.
* Gender: Both male and female patients will be included.
* Patients have established diagnosis of NASH (based on liver ultrasonography).

Exclusion Criteria:

* Young ages <18 years
* Secondary causes of hepatic fat accumulation such as Significant alcohol consumption as defined by an average daily consumption of alcohol greater than 30 g/day in men and greater than 20 g/day in women or Long-term use of a steatogenic medication (e.g., non-Steroidal anti-inflammatory drugs (NSAIDs) amiodarone, methotrexate, tamoxifen, corticosteroids)
* Patients with a known history of viral hepatitis, hemochromatosis, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, biliary obstruction.
* Patients with inflammatory diseases.
* Subjects using any other lipid-lowering agents, or any supplements known to have antioxidant activity and omega-3 supplementation for at least 3 months before participation in the trial
* Current Pregnancy
* Breastfeeding
* Females On Oral Contraceptive pills
* Patients with renal impairment
* Patients with heart failure
* Patients with cancer or with a history of cancer treatment
* Any contraindications to coenzyme Q 10 Or statins like hypersensitivity to anyone
* Patients with predisposing risk factors for myopathy/rhabdomyolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness measurement (LSM) | At baseline and 12th week
  LSM will be assessed by Fibro scan
Change in ultrasound score | At baseline and 12th week
  Ultrasound score will be assessed by Ultrasonography

SECONDARY OUTCOMES:
Demonstrate changes in Alanine aminotransferase (ALT) | At baseline and 12th week
  Alanine aminotransferase (ALT) in U/L
Demonstrate changes in Aspartate aminotransferase (AST) | At baseline and 12th week
  Aspartate aminotransferase (AST) in U/L
Demonstrate changes in Alkaline phosphatase (ALP) | At baseline and 12th week
  Alkaline phosphatase (ALP) in U/L
Demonstrate changes in ɤ-glutamyltranspeptidase (GGT) | At baseline and 12th week
  ɤ-glutamyltranspeptidase (GGT) in U/L
Demonstrate changes in Direct bilirubin | At baseline and 12th week
  Direct bilirubin in mg/dl
Demonstrate changes in the Lipid values | At baseline and 12th week
  Total cholesterol(TC) in mg/dl , Triglycerides(TG) in mg/dl , LDL-Cholesterol in mg/dl , HDL-Cholesterol in mg/dl
Demonstrate changes in the body weight and body mass index (BMI) | At baseline and 12th week
  BMI in kg/m^2 will be calculated using the formula: BMI= [Weight (kg)/Height (m2)].
Demonstrate changes in the Inflammatory marker : CRP | At baseline and 12th week
  C-reactive protein in mg/L
Demonstrate changes in Serum cytokeratin 18 (Ck-18) | At baseline and 12th week
  Serum cytokeratin 18 (Ck-18) will be determined by Enzyme-linked Immunosorbent assay kits.
Demonstrate changes in Serum transforming growth factor-beta1 (TGF-β1) | At baseline and 12th week
  Serum transforming growth factor-beta1 (TGF-β1) will be determined by Enzyme-linked Immunosorbent assay kits.
Serum Retinol binding protein 4 (RBP-4) | At baseline and 12th week
  Serum Retinol binding protein 4 (RBP-4) will be determined by Enzyme-linked Immunosorbent assay kits.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer Ahmed Alsayed, B.Sc. Degree, Principal Investigator — Faculty of pharmacy , Pharos University

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Estes C, Anstee QM, Arias-Loste MT, Bantel H, Bellentani S, Caballeria J, Colombo M, Craxi A, Crespo J, Day CP, Eguchi Y, Geier A, Kondili LA, Kroy DC, Lazarus JV, Loomba R, Manns MP, Marchesini G, Nakajima A, Negro F, Petta S, Ratziu V, Romero-Gomez M, Sanyal A, Schattenberg JM, Tacke F, Tanaka J, Trautwein C, Wei L, Zeuzem S, Razavi H. Modeling NAFLD disease burden in China, France, Germany, Italy, Japan, Spain, United Kingdom, and United States for the period 2016-2030. J Hepatol. 2018 Oct;69(4):896-904. doi: 10.1016/j.jhep.2018.05.036. Epub 2018 Jun 8. PMID 29886156
- [Background] Mantovani A, Scorletti E, Mosca A, Alisi A, Byrne CD, Targher G. Complications, morbidity and mortality of nonalcoholic fatty liver disease. Metabolism. 2020 Oct;111S:154170. doi: 10.1016/j.metabol.2020.154170. Epub 2020 Jan 30. PMID 32006558
- [Background] Ekstedt M, Hagstrom H, Nasr P, Fredrikson M, Stal P, Kechagias S, Hultcrantz R. Fibrosis stage is the strongest predictor for disease-specific mortality in NAFLD after up to 33 years of follow-up. Hepatology. 2015 May;61(5):1547-54. doi: 10.1002/hep.27368. Epub 2015 Mar 23. PMID 25125077
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Vanni E, Marengo A, Mezzabotta L, Bugianesi E. Systemic Complications of Nonalcoholic Fatty Liver Disease: When the Liver Is Not an Innocent Bystander. Semin Liver Dis. 2015 Aug;35(3):236-49. doi: 10.1055/s-0035-1562944. Epub 2015 Sep 17. PMID 26378641
- [Background] Spahillari A, Mukamal KJ, DeFilippi C, Kizer JR, Gottdiener JS, Djousse L, Lyles MF, Bartz TM, Murthy VL, Shah RV. The association of lean and fat mass with all-cause mortality in older adults: The Cardiovascular Health Study. Nutr Metab Cardiovasc Dis. 2016 Nov;26(11):1039-1047. doi: 10.1016/j.numecd.2016.06.011. Epub 2016 Jun 28. PMID 27484755
- [Background] Tzanaki I, Agouridis AP, Kostapanos MS. Is there a role of lipid-lowering therapies in the management of fatty liver disease? World J Hepatol. 2022 Jan 27;14(1):119-139. doi: 10.4254/wjh.v14.i1.119. PMID 35126843
- [Background] Wang W, Zhao C, Zhou J, Zhen Z, Wang Y, Shen C. Simvastatin ameliorates liver fibrosis via mediating nitric oxide synthase in rats with non-alcoholic steatohepatitis-related liver fibrosis. PLoS One. 2013 Oct 2;8(10):e76538. doi: 10.1371/journal.pone.0076538. eCollection 2013. PMID 24098525
- [Background] Pramfalk C, Parini P, Gustafsson U, Sahlin S, Eriksson M. Effects of high-dose statin on the human hepatic expression of genes involved in carbohydrate and triglyceride metabolism. J Intern Med. 2011 Mar;269(3):333-9. doi: 10.1111/j.1365-2796.2010.02305.x. Epub 2010 Nov 18. PMID 21083855
- [Background] Farsi F, Mohammadshahi M, Alavinejad P, Rezazadeh A, Zarei M, Engali KA. Functions of Coenzyme Q10 Supplementation on Liver Enzymes, Markers of Systemic Inflammation, and Adipokines in Patients Affected by Nonalcoholic Fatty Liver Disease: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial. J Am Coll Nutr. 2016 May-Jun;35(4):346-53. doi: 10.1080/07315724.2015.1021057. Epub 2015 Jul 9. PMID 26156412
- [Background] Chen K , Chen X , Xue H , Zhang P , Fang W , Chen X , Ling W . Coenzyme Q10 attenuates high-fat diet-induced non-alcoholic fatty liver disease through activation of the AMPK pathway. Food Funct. 2019 Feb 20;10(2):814-823. doi: 10.1039/c8fo01236a. PMID 30675881